CLINICAL TRIAL: NCT06867887
Title: Non-invasive Detection of Driveline Infections in Patients with a Left Ventricular Assist Device
Acronym: DRIVE-ID
Status: Enrolling by invitation | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, Kadir Caliskan MD, PhD, FESC, Cardiologist, Erasmus Medical Center
Other Study IDs: MEC-2023-0597
Record Dates: First submitted 2024-09-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-09

CONDITIONS: LVAD (Left Ventricular Assist Device) Driveline Infection
Keywords: Infection; LVAD; Detection; Monitoring; Driveline infection; Imaging; Non-invasive
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients implanted with an LVAD

SUMMARY:
The aim of this single center observational study is to determine the feasibility of using non-invasive imaging methods, including smartphone photography and infrared thermography, for detecting of DLIs in LVAD patients in terms of severity, extent and natural healing process.

DETAILED DESCRIPTION:
Observational data of the driveline exit of LVAD patients will be collected during a follow-up period of 26 weeks. Two non-invasive imaging methods will be used.

Smartphone photos will be taken weekly by the patient during routine wound care in the home environment.

In case the patient is admitted for driveline infection, infrared thermographic (IRT) photography will be used to make thermographic photos of the driveline exit and the abdominal area of the subcutaneous driveline.

Furthermore, existing smartphone images and diagnostic data regarding prior DLI status will be obtained from the electronic patient records.

Imaging data will additionally be retrospectively analyzed using artificial intelligence (AI) and machine learning for the development of a predictive AI model.

ELIGIBILITY:
Inclusion Criteria: Patients age 16 years or older, implanted with an LVAD, followed at Erasmus MC, with access to a smartphone with a built-in camera, who have signed an informed consent for data collection.

Exclusion Criteria: Known cognitive problems, like dementia etc., non-cardiac disease or cardiac diseases resulting in a life expectancy less than 1 years, inability to read or sign the informed consent form.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with an LVAD
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Extent and severity of driveline infections in LVAD patients using non-invasive imaging | 26 weeks
  Assess the extent, severity, and healing process of LVAD driveline infections in patients on LVAD support
Driveline exit healing process and risk of infection of the LVAD driveline | 26
  Assess the healing process of the driveline exit using non-invasive imaging (smartphone and thermographic)

SECONDARY OUTCOMES:
Sceptic complications | 26 weeks
  Occurance of systemic infection, positive blood cultures, and VAD-related infections.
Machine learning model for predicting DLIs. | 26 weeks
  Assess whether a machine learning model can be developed and validated based on smartphone photography and IRT to predict the occurrence of DLIs.

CONTACTS AND LOCATIONS:
Overall Officials: K. Caliskan, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Imaging data will be de-identified and then shared with Eindhoven University of Technology for further analyses and modeling.
Supporting Information: Study Protocol
Time Frame: Data transfer is anticipated 1 October 2024 and 1 July 2025
Access Criteria: Coordinating researcher V. Drost will be able to access the IPD and supporting information via the investigation site.